CLINICAL TRIAL: NCT03665792
Title: The Prospective Observational Research of the Analgesic Effect of Sevoflurane and the Correlation Between Sevoflurane and qNOX
Brief Title: The Correlation Between Sevoflurane and qNOX
Status: Completed | Type: Observational
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Other Study IDs: CINI-ZYLX-201806-11
Record Dates: First submitted 2018-08-04; First posted 2018-09-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Analgesic Adverse Reaction; Nociceptive Pain; Inhalation; Vapor
MeSH Terms: conditions — Nociceptive Pain; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: nociception index qNOX — non-invasive, real time, monitoring for nociception stimulation
  Other Names: CON , BIS

SUMMARY:
This study purpose to observation the sevoflurane analgesia effect, and using nociception real-time monitoring NOX to test the correlation between the sevoflurane and NOX index.

DETAILED DESCRIPTION:
This study purpose to observation the sevoflurane analgesia effect, and using nociception real-time monitoring NOX to test the analgesia effect of the sevoflurane.

And test the correlation between the sevoflurane and NOX index.

ELIGIBILITY:
Inclusion Criteria:

1. Elective thoracoscope surgery patients
2. Age ranging from 25 to 85 years
3. American Society of Anesthesiologists (ASA) Physical Status score of 2 to 4
4. a body mass index (BMI) ranging from 18.5 to 40 kg/m2.

Exclusion Criteria:

1. Clinical diagnosis of Alzheimer's Disease
2. implanted pacemaker
3. Clinical diagnosis of psychiatric diseases
4. Clinical diagnosis of epilepsy
5. Clinical diagnosis of autonomic nervous system disorders which might affect the EEG

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: only elective thoracoscope surgery patients were enrolled
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The sevoflurane application correlated with the qNOX index | through study completion, an average of 1 year
  The sevoflurane application correlated with the qNOX index, meanwhile reflect the analgesia effect of sevoflurane application

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wang, MD,PHD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Bei Liu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No